CLINICAL TRIAL: NCT06823856
Title: Open-label, Randomized, Two-period Comparative Pharmacokinetics and Bioequivalence Study of Empagliflozin + Metformin Hydrochloride 12.5 mg/1000 mg Film-coated Tablets (Gedeon Richter Plc., Hungary) Versus Synjardy 12.5 mg/1000 mg Film-coated Tablets (Boehringer Ingelheim International GmbH, Germany) in Healthy Volunteers Under Fed Conditions
Brief Title: Pharmacokinetics and Bioequivalence Study of Empagliflozin+Metformin Hydrochloride 12.5 mg/1000 mg Film-coated Tablets (Gedeon Richter Plc., Hungary) Versus Synjardy 12.5 mg/1000 mg Film-coated Tablets (Boehringer Ingelheim International GmbH, Germany)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: EAEU-GCO-MET/EMP-03-2023
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: Diabetes; Diabetes Mellitus Type 2; Empagliflozin; Metformin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — empagliflozin; Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Empagliflozin + Metformin hydrochloride combination film-coated tablets (Experimental): Combination tablet of Empagliflozin + Metformin hydrochloride 12.5 mg/1000 mg of Gedeon Richter Plc., Hungary
  Interventions: Drug: Empagliflozin + Metformin hydrochloride 12.5 mg/1000 mg combination film-coated tablets
- Synjardy film-coated tablets (Active Comparator): Synjardy 12.5 mg/1000 mg of Boehringer Ingelheim International GmbH, Germany
  Interventions: Drug: Synjardy 12.5 mg/1000 mg film-coated tablets

INTERVENTIONS:
Drug: Empagliflozin + Metformin hydrochloride 12.5 mg/1000 mg combination film-coated tablets — 1 tablet of Empagliflozin + Metformin hydrochloride 12.5 mg/1000 mg combination film-coated table
  Arms: Empagliflozin + Metformin hydrochloride combination film-coated tablets
Drug: Synjardy 12.5 mg/1000 mg film-coated tablets — 1 tablet of Empagliflozin+Metformin 12.5 mg/1000 mg filmcoated tablets
  Arms: Synjardy film-coated tablets

SUMMARY:
Empagliflozin and metformin hydrochloride are two separate drugs. The combination of these two drugs in one tablet are used for the treatment of type 2 diabetes, along with diet and exercise, and can be used with other drugs, if required. It is approved in Russia and also various other countries. In Russia, the brand name is Synjardy®.

The purpose of this research study is to measure the amount of the two drugs in the blood after taking two different formulations of the combination tablet. One formulation, also called Synjardy®, is an approved product in Russia marketed by Boehringer Ingelheim International GmbH, Germany. The other formulation is an investigational product that is not approved. The data from this study will be used to compare the two products.

Subjects participating in this study will take 12.5 mg empagliflozin and 1000 mg metformin hydrochloride (1 combination film-coated tablet) of one formulation in each period. The maximum recommended daily dose is 25 mg of empagliflozin and 2,000 mg of metformin hydrochloride which is based on the subject's current regimen, effectiveness, and tolerability.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of the written informed consent of the volunteer to participate in the study in accordance with the current legislation, volunteer's agreement to observe all study restrictions and consent to come back to the center for providing of all study procedures.
2. Verified as "healthy" by the Investigator based on the results of the standard clinical and laboratory tests and instrumental investigations, results of physical examination and medical history data;
3. Male and female volunteers of Caucasian race, aged 18 to 45 years (inclusive) at screening.

   Female volunteers can be with childbearing or non-childbearing potential. Female volunteers of non-childbearing potential are defined as: females with documented menopause (defined as the absence of menstruation for at least 12 consecutive months without an alternative medical cause with follicle-stimulating hormone (FSH) level at screening ≥25 mIU/mL) or females with documented surgical sterilization (hysterectomy, bilateral ovary- or tubectomy, uterine tubes ligation);
4. Body mass index (BMI) (by Quetelet) between 18.5 and 30 kg/m2 (inclusive). Body weight must be more than 45 kg and less than 100 kg;
5. A volunteer must agree the following requirements:

   1. Female volunteers of childbearing potential must confirm the absence of unprotected sexual intercourse with unsterilized partner within 30 days before screening;
   2. Female volunteers must agree to sexual abstinence or to use consistently and correctly one of the adequate contraceptive methods listed below during their participation in this study and for 30 days after the last dose of the IMP;
   3. Male volunteers must agree to sexual abstinence or together with their female partners of childbearing potential must use consistently and correctly one of the adequate contraceptive methods listed below during their participation in this study and for 30 days after the last dose of the IMP;
   4. Male volunteers must agree to refrain from donating sperm during their participation in this study and for 30 days after the last dose of the IMP;

   Note: Adequate contraceptive methods include:
   * Non-hormonal intrauterine device (IUD);
   * Barrier method in combination with spermicidal drug or diaphragm (diaphragm with spermicide, cervical cap with spermicide, condom with spermicide).
6. A volunteer has suitable veins for cannulation.

Exclusion Criteria:

1. Known history or presence of clinically significant neurologic, hematologic, endocrine (including diabetes mellitus 1 and 2 type), oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results;
2. Known history or presence of clinically significant disease of the gastrointestinal tract, surgical interventions on gastrointestinal tract (except appendectomy);
3. Burdened allergological anamnesis, including known history of anaphylactic reaction/anaphylactic shock, known history or presence of hypersensitivity or idiosyncratic reaction to empagliflozin or metformin or excipients of the test/reference product, or any other drug substances with similar activity;
4. Acute or chronic infectious disease within 4 weeks before screening;
5. History or presence of malignant disease;
6. Presence of clinically significant hepatic or renal dysfunction as per Investigator's discretion;
7. Estimated creatinine clearance of ≤60 mL/min based on the Cockcroft-Gault equation, or serum creatinine level higher than the upper limit of normal range of the local laboratory;
8. Use of medication (prescribed, over-the-counter medications, and natural health products [including herbal remedies, phytohormones, homeopathic and traditional medicines, probiotics, food supplements such as vitamins, minerals, amino acids, essential fatty acids, and protein supplements used in sports]) within 14 days prior to screening and thereafter. It is allowed to use medical products without systemic absorption.
9. Use of medications with potent effect on hemodynamics, and liver function (barbiturates, omeprazole, cimetidine, etc.) within 30 days before screening and thereafter;
10. Donation of blood or plasma (450 ml and more) within 2 months before screening;
11. Blood or plasma transfusion within 1 year before screening;
12. Results of standard laboratory investigations outside the normal range of the local laboratory, which are considered clinically significant by the Investigator;
13. ECG abnormalities, including clinically significant arrhythmia, or suspected arrhythmia as judged by the Investigator;
14. Vital sign abnormalities at the screening (systolic blood pressure [BP] < 100 or > 130 mmHg, diastolic BP < 60 or > 90 mmHg, or heart rate [HR] < 60 or > 90 bpm);
15. Positive test for hepatitis B, hepatitis C, human immunodeficiency virus (HIV), or syphilis. It is allowed to use results of the HIV test, hepatitis viruses B and C tests and syphilis analysis, which were performed within 3 months before screening visit;
16. Positive test for SARS-CoV-2 using express immunochromatographic test system for qualitative detection of SARS-CoV-2 antigen in smears from the nasopharynx or oropharynx;
17. Positive urine cotinine test at screening or at Day 0, or smoking cigarettes or tobacco or consuming any nicotine products (patches, chewing gum etc.) during 6 months prior to screening;
18. Positive alcohol breath test at screening or at Day 0, or history of significant alcohol abuse within one year prior to screening, regular use of alcohol within 6 months prior to screening (more than 10 units of alcohol per week [1 unit = 200 mL of dry wine, 400 mL of beer, or 50 mL of 40% alcohol]), or consumption of alcohol within 72 hours prior to screening/72 hours prior to dosing;
19. Positive urine screening for narcotic, psychotropic, and potent substances at screening or at Day 0, or history of significant drug abuse or use of illegal drugs (such as marijuana, cocaine, phencyclidine, crack, opioid derivatives including heroin, and amphetamine derivatives).
20. Positive pregnancy test at screening or at Day 0 (the test is performed to all female volunteers);
21. Female volunteers who are pregnant or lactating, who wish to get pregnant; female volunteers of childbearing potential with presence of unprotected sexual intercourse with unsterilized partner within 30 days before screening; male subjects who wish to conceive during participation in the study;
22. Female volunteers who have used hormonal contraceptives (implanted, injected, intravaginal, or intrauterine hormonal contraceptives within 6 months prior to screening; oral or transdermal hormonal contraceptives within 21 days prior to screening) or wish to use them during participation in the study;
23. Consumption of food containing poppy seeds within 72 hours prior screening / 72 hours prior to hospitalization in the first period;
24. Consumption of food or beverages containing xanthine derivatives or xanthine-related compounds (e.g. tea, coffee, cola, chocolates) or energy drinks from 72 hours prior to first dosing;
25. Consumption of food or beverages containing grapefruit, starfruit, pomegranate, pineapple, or pomelo from 14 days prior to the first dosing;
26. Dehydration due to diarrhea, vomiting or other causes during the last 24 hours before dosing;
27. Participation in a clinical trial that involved administration of an investigational medicinal product within 30 days prior to drug administration or within 5 times the half-life of the previous IMP used, whichever is longer, or recent participation in a clinical investigation that, in the opinion of the Investigator, would jeopardize subject safety or the integrity of the study results;
28. Difficulties with staying fasting or consuming standardized high-calorie breakfast/other meal provided by the site;
29. Planned or scheduled surgery within 7 days prior or 7 days after study drugs administration;
30. Difficulties with swallowing tablets or capsules whole;
31. Following a special diet within 30 days prior to the first drug administration (e.g., liquid, protein, raw food diet, vegetarian, vegan);
32. Mental, physical or other reasons that do not allow the volunteer to adequately assess his/her behaviour and correctly fulfil the conditions of the study protocol;
33. Other diseases/conditions that, in the opinion of the Investigator, may affect the pharmacokinetics of the study drugs or increase the risk for the health of the volunteer;
34. Any reason which, in the opinion of the Investigator, would prevent the volunteer from participating in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2025-05-11 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-05-21 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of Empagliflozin + Metformin hydrochloride film-coated tablets and Synjardy® film-coated tablets via measuring the AUC from time 0 to last collection time t (AUC0-t) | From enrollment to the end of treatment at about 7 weeks
  The primary purpose of the study is to assess the bioequivalence of Empagliflozin + Metformin hydrochloride 12.5 mg/1000 mg film-coated tablets (Gedeon Richter Plc., Hungary) and Synjardy 12.5 mg/1000 mg film-coated tablets (Boehringer Ingelheim International GmbH, Germany) in healthy, adult volunteers under fed conditions. The measurement will be based on two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data of AUC.
Bioequivalence of Empagliflozin + Metformin hydrochloride film-coated tablets and Synjardy® film-coated tablets via measuring the maximum concentration in plasma (Cmax) | From enrollment to the end of treatment at about 7 weeks
  The primary purpose of the study is to assess the bioequivalence of Empagliflozin + Metformin hydrochloride 12.5 mg/1000 mg film-coated tablets (Gedeon Richter Plc., Hungary) and Synjardy 12.5 mg/1000 mg film-coated tablets (Boehringer Ingelheim International GmbH, Germany) in healthy, adult volunteers under fed conditions. The measurement will be based on two-sided 90% CI for the test to reference ratio of the population means is within 80.00% to 125.00% for each of the Ln-transformed data of Cmax.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From enrollment to the end of treatment at about 7 weeks
  The secondary purpose is to assess the safety and tolerability of the study products from the signing of the informed consent form (ICF) until the end of the study. There will be no formal statistical evaluation of safety or tolerability. The safety results will be provided as listings and summary tables for each treatment group. Adverse event data listing will include AEs onset and resolution date/time, duration, time from dosing, severity, relationship to the IMP and/or the additional drug product, outcome, and the action taken to the IMP and/or additional drug product and to treat the AE.

CONTACTS AND LOCATIONS:
Locations (1):
- State Budgetary Institution of Healthcare of Yaroslavl region "Yaroslavl Regional Clinical Narcological Hospital, Yaroslavl, Russia

IPD SHARING:
Plan to Share IPD: No